CLINICAL TRIAL: NCT03571880
Title: Intra- And Inter-operator Reliability Of Isometric Back And Abdominal Muscle Strength Testing In Healthy Controls And Persons With Nonspecific Chronic Low Back Pain.
Acronym: LBP-BIO-REL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LBP-BIO-REL-001
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CNSLBP group (Experimental)
  Interventions: Device: Biodex-assisted isometric strength testing
- Healthy control group (Active Comparator)
  Interventions: Device: Biodex-assisted isometric strength testing

INTERVENTIONS:
Device: Biodex-assisted isometric strength testing — The maximum voluntary isometric and dynamic strength of back and abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).

SUMMARY:
Low back pain (LBP) is currently the most common cause of functional impairment with regard to the musculoskeletal system1. LBP occurs in men and women in all age groups and has a peak incidence between 30 and 65 years. Although 10% of the persons with LRP can be diagnosed with a specific underlying pathology (e.g., disc herniation, canal stenosis, spondylolysis, ...), 90% have symptoms with an unclear origin. 23% of the latter group will eventually develop chronic nonspecific low back pain (CNSLBP)2.

Exercise therapy is seen as an important component in the rehabilitation of persons with CNSPLBP3. Because previous research showed reduced muscle strength of the back muscles4, exercise therapy that improves / recovers muscle strength is being investigated. However, there is still a lack of clarity concerning the effect that reduced muscle strength has on the development and further development of back pain5-6. The objective testing of back muscle strength remains a recurring issue. Up to now, back muscle strength has been mainly tested by a battery of clinical tests (eg Sorensen test) or the use of "iso machines"7. These Iso machines contain a dynamometer that can very specifically reflect the isometric or isokinetic force on an axis of rotation. Different types of these iso machines (eg Cybex, Biodex) have already been developed, each with specific designs (eg differences in the hip angle, differences in the stabilization of the participant). However, to date no standardized protocols are available for evaluating both abdominal and back muscle strength. Furthermore, it is also essential that before such systems can be used in clinical intervention studies, the reliability of such systems is investigated and that reference data from healthy subjects are collected with which data from patients can be compared.

The aim of the current research is therefore to investigate the intra- and inter-operator reliability of a standardized protocol drawn up according to the latest scientific evidence. A second goal is to set standard values for healthy persons for the developed protocol using the Biodex 3 dynamometer system.

ELIGIBILITY:
Inclusion Criteria:

1. medically diagnosed with non-specific chronic low back pain,
2. between 25-60 years old,
3. able to understand Dutch (spoken and written).

Exclusion Criteria:

1. invasive surgery at the lumbar spine in the last 18 months (arthrodesis was excluded, microsurgery was allowed),
2. radiculopathy (uni- or bilateral),
3. co-morbidities: paresis and/or sensory disturbances by neurological causes, diabetes mellitus, rheumatoid arthritis, pregnancy,
4. ongoing compensation claims and/or (work)disability > 6 months,
5. rehabilitation/exercise therapy program for LBP in the past 6 months.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
abdominal isometric strength | day1
  The maximum voluntary isometric strength of the abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Abdominal isometric strength | day 2
  The maximum voluntary isometric strength of the abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Abdominal dynamic strength | day 1
  The maximum voluntary dynamic strength of abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Abdominal dynamic strength | day 2
  The maximum voluntary dynamic strength of abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Back isometric strength | day 1
  The maximum voluntary isometric strength of the back muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Back isometric strength | day 2
  The maximum voluntary isometric strength of the back muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Back dynamic strength | day 1
  The maximum voluntary dynamic strength of back muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Back dynamic strength | day 2
  The maximum voluntary dynamic strength of back muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).

SECONDARY OUTCOMES:
Pain | day 1
  The Numeric Pain Rating Scale (NPRS) is a nominal scale on which the participant indicates the amount of pain he/she perceives at that current moment. It consists of a line indicating eleven successive scores (0-10), whereby score 0 means 'no pain' and score 10 means 'worst pain imaginable'. An improvement of 2 levels or more is accepted as clinically relevant.
The Modified Oswestry Disability Index (ODI) | Day 1
  The Modified Oswestry Disability Index (ODI) is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of 10 items that are scored on a 5-point scale. The total score gives a percentage degree of limitation for the patient.
Physical Activities Scale For Individuals with Physical Disabilities (PASIPD) | day 1
  The PASIPD is a questionnaire consisting of 13 items to measure the physical activity of people with disabilities. It provides information about leisure, household and work-related physical activity in the last 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Verbrugghe, drs, Study Chair — Hasselt University; Annick Timmermans, prof. dr., Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt
  - Jessa Ziekenhuis, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Result] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Result] van Middelkoop M, Rubinstein SM, Kuijpers T, Verhagen AP, Ostelo R, Koes BW, van Tulder MW. A systematic review on the effectiveness of physical and rehabilitation interventions for chronic non-specific low back pain. Eur Spine J. 2011 Jan;20(1):19-39. doi: 10.1007/s00586-010-1518-3. Epub 2010 Jul 18. PMID 20640863